CLINICAL TRIAL: NCT06401083
Title: The Effect of an Additional Pre-extubational Loading Dose of Caffeine-citrate
Acronym: NEOKOFF22
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Semmelweis University (Other)
Responsible Party: Principal Investigator, Dr. Gasparics Ákos, Chief Investigator, Assistant Lecturer, Semmelweis University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NEOKOFF22; 2022-003202-77 (EudraCT Number)
Record Dates: First submitted 2024-03-18; First posted 2024-05-06 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-04

CONDITIONS: Apnea of Prematurity; Premature Birth; Respiratory Failure
Keywords: prematurity; caffeine; methylxanthine; apnea of prematurity; extubation failure
MeSH Terms: conditions — Apnea; Premature Birth; Respiratory Insufficiency | interventions — caffeine citrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre-extubational caffeine-citrate (Active Comparator): Participants will receive 20 mg/kg loading dose of caffeine citrate on the first day of life and after that 5-10 mg/kg maintenance dose each day. On this arm, the participants will receive 20 mg/kg caffeine dose once again before the planned extubation.
  Interventions: Drug: Caffeine citrate
- Routine care (No Intervention): Participants will receive 20 mg/kg loading dose of caffeine citrate on the first day of life and after that 5-10 mg/kg maintenance dose each day, also on the day of the extubation.

INTERVENTIONS:
Drug: Caffeine citrate — 20 mg/kg caffeine-citrate before the planned extubation.
  Other Names: CITRATE DE CAFEINE COOPER 25 mg/ml Coopération Pharmaceutique Française, Melun, France
  Arms: Pre-extubational caffeine-citrate

SUMMARY:
The goal of this clinical trial is to answer whether the use of a single loading dose (20 mg/kg) of caffeine citrate one hour before extubation has an impact on the success rate of extubation among preterm neonates. In addition, the investigators would like to assess the frequency of apneas and side effects of the intervention, as well as the development of NEC, BPD, IVH, PVL, and long-term neurodevelopmental outcomes in the investigated populations.

According to institutional protocol, preterm infants born before the 32nd week of gestation receive a standard dose of caffeine citrate therapy. This covers a maintenance dose of 5-10 mg/kg of caffeine citrate administered intravenously once or twice daily after a loading dose of 20 mg/kg on the first day of life. In this trial, preterm infants born before the 32nd gestational week and who had been mechanically ventilated for at least 48 hours before planned extubation are planned to be randomly allocated into intervention and control groups. The intervention group will receive an additional loading dose of caffeine citrate 60 minutes before extubation. The control group will receive standard dosing regimens.

DETAILED DESCRIPTION:
The most common cause of the failure of non-invasive ventilatory support is poor spontaneous respiratory activity in preterm infants and recurrent respiratory arrest (apnea) due to the immature nervous system. The national and international literature has extensively studied apnea in preterm infants. Apnea is a respiratory failure of 15-20 seconds or shorter duration associated with bradycardia or desaturation. Apneas develop in preterm infants due to prematurity of the respiratory center and chemoreceptors and reduced patency of the upper airway. Apnea in preterm infants is the most common indication for intubation and reintubation.

The apnea-reducing effects of the respiratory center stimulant methylxanthines have been known for more than 40 years. Based on current knowledge, caffeine is the drug of choice for the medical treatment of apnea. Caffeine has the narrowest spectrum of side effects, the broadest therapeutic range, and the most prolonged half-life among methylxanthines.

Caffeine is currently one of the most commonly used drugs in premature neonatal intensive care units. The most common dosing recommendation is a maintenance dose of 5-10 mg/kg daily after a loading dose of 20 mg/kg of caffeine citrate. Higher saturating and maintenance doses have been used in some studies, with some reports suggesting that higher doses of caffeine increase the chance of successful extubation. However, other studies have reported more frequent adverse effects at higher doses. Conflicting literature suggests that caffeine dosing may vary between institutions. Further basic research and clinical studies are needed to determine the optimal dose.

The investigators seek to answer whether the use of a single loading dose of caffeine citrate one hour before extubation impacts the success rate of extubation. In addition, the investigators would like to assess the frequency and severity of side effects and the development of necrotizing enterocolitis, intraventricular hemorrhage, periventricular leukomalacia, and bronchopulmonary dysplasia.

To investigate the effect of a pre-extubational loading dose of caffeine-citrate, the investigators plan to carry out a two-armed randomized clinical trial, including preterm neonates being treated in one of the tertiary neonatal intensive care units of Semmelweis University. A total of 226 patients are planned to be enrolled. According to institutional protocol, preterm infants born before the 32nd week of gestation receive a standard dose of caffeine therapy. This covers a maintenance dose of 5-10 mg/kg of caffeine citrate administered intravenously once or twice daily after a loading dose of 20 mg/kg on the first day of life.

Preterm infants who have been on mechanical ventilation for at least 48 hours before planned extubation will be randomly allocated into intervention and control groups. Stratification of the randomization will be based on gestational age and antenatal steroid prophylaxis. Intervention is an additional loading dose (20 mg/kg) of intravenous caffeine citrate 60 minutes before extubation. The control group will receive routine dosing regimens as mentioned above. Before extubation, the parents will be informed and asked for consent. Pre-interventional, the investigators plan to collect baseline characteristics and oxygen requirements. After extubation, the need for reintubation within the next 48 hours will be assessed. This timeframe was chosen because most of reintubation due to respiratory reasons happens within the next 48 hours after extubation, and the caffeine half-life ranges from 40 to 230 hours.

The investigators will also assess the frequency of side effects such as gastric residuals, frequency of apneas, need for supplementary oxygen, elevated heart rate, or blood pressure. Data will be collected about adverse outcomes of prematurity, e.g., necrotizing enterocolitis, intraventricular hemorrhage, periventricular leukomalacia, and bronchopulmonary dysplasia.

ELIGIBILITY:
Inclusion Criteria:

* Premature infant born before 32nd week of gestation is completed;
* Had been mechanically ventilated for at least 48 hours;
* Before the first planned extubation.

Exclusion Criteria:

* Lack of informed consent, refusal to participate in the study;
* Major congenital anomaly;
* Had not received surfactant treatment;
* Hydrops foetalis;
* Persistent tachycardia before extubation, fetal/neonatal arrhythmia;
* Asphyxia.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 226 (Estimated)
Dates: Start 2023-12-21 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Rate of extubation failure | 48 hours
  Reintubation. The discretion of the attending physician.

SECONDARY OUTCOMES:
Frequency of apneas | 48 hours
  Respiratory failure of 15-20 seconds or shorter duration associated with bradycardia or desaturation.
Change in the mean heart rate | 72 hours
  Mean heart rate measured 24 hours before and 48 hours after intervention.
Tachycardia | 72 hours
  The time interval when the heart rate >200 (min) during one day (1440 min) in percentage.
Volume of gastric residuals | 72 hours
  Gastric residuals measured 24 hours before and 48 hours after intervention.
Reduction/Cessation of feeding | 48hours
  48 hours after intervention.
Change in mean arterial blood pressure | 48 hours
  Mean blood pressure measured 24 hours before and after intervention measured with non-invasive methods.
Mechanical ventilation (MV) days | At discharge from participating centres, an average of one month.
  MV days during the length of hospital stay
Non-invasive ventilation (NIV) days | At discharge from participating centres, an average of one month.
  NIV days during the length of hospital stay
Rate of necrotizing enterocolitis | At discharge from participating centres, an average of one month.
  Development of necrotizing enterocolitis according to Bell stages.
Rate of Intraventricular hemorrhage | At discharge from participating centres, an average of one month.
  Development or progression of intraventricular hemorrhage according to Papile stages diagnosed with cranial ultrasound.
Rate of periventricular leukomalacia | At discharge from participating centres, an average of one month.
  Development of periventricular leukomalacia, seen on cranial ultrasound.
Rate of late-onset sepsis | At discharge from participating centres, an average of one month.
  Culture proven sepsis after the first 72 hours of life.
Rate of patent ductus arteriosus | At discharge from participating centres, an average of one month.
  Pharmacological or surgical treatment was required.
Rate of bronchopulmonary dysplasia | 36th postmenstrual age
  Diagnosis of bronchopulmonary dysplasia.
Rate of death before discharge | At discharge from participating centres, an average of one month.
Required oxygen concentration | 24 hours
  Required oxygen concentration before and after the intervention.
Long term neurodevelopmental outcome | At 2 years of corrected age
  Measured by Bayley score. The standardized mean score is 100 (SD 15), with scores lower than 85 indicating mild impairment, and lower than 70 indicating moderate or severe impairment.
Severity of sensoric or motoric impairment | At 2 years of corrected age
  Hearing or visual impairment, and cerebral palsy

CONTACTS AND LOCATIONS:
Overall Officials: Ákos Gasparics, MD.PhD, Principal Investigator — Semmelweis University, Department of Obstetrics and Gynecology
Locations (2):
- Hungary (2):
  - Pediatric Center, Semmelweis University, Budapest
  - Department of Obstetrics and Gynecology, Semmelweis University, Budapest

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Erickson G, Dobson NR, Hunt CE. Immature control of breathing and apnea of prematurity: the known and unknown. J Perinatol. 2021 Sep;41(9):2111-2123. doi: 10.1038/s41372-021-01010-z. Epub 2021 Mar 12. PMID 33712716
- [Background] Bacci SLLDS, Johnston C, Hattori WT, Pereira JM, Azevedo VMGO. Mechanical ventilation weaning practices in neonatal and pediatric ICUs in Brazil: the Weaning Survey-Brazil. J Bras Pneumol. 2020 Mar 23;46(4):e20190005. doi: 10.36416/1806-3756/e20190005. eCollection 2020. PMID 32215452
- [Background] Kreutzer K, Bassler D. Caffeine for apnea of prematurity: a neonatal success story. Neonatology. 2014;105(4):332-6. doi: 10.1159/000360647. Epub 2014 May 30. PMID 24931325
- [Background] Schmidt B, Roberts RS, Davis P, Doyle LW, Barrington KJ, Ohlsson A, Solimano A, Tin W; Caffeine for Apnea of Prematurity Trial Group. Caffeine therapy for apnea of prematurity. N Engl J Med. 2006 May 18;354(20):2112-21. doi: 10.1056/NEJMoa054065. PMID 16707748
- [Background] Schmidt B, Roberts RS, Davis P, Doyle LW, Barrington KJ, Ohlsson A, Solimano A, Tin W; Caffeine for Apnea of Prematurity Trial Group. Long-term effects of caffeine therapy for apnea of prematurity. N Engl J Med. 2007 Nov 8;357(19):1893-902. doi: 10.1056/NEJMoa073679. PMID 17989382
- [Background] Eichenwald EC. National and international guidelines for neonatal caffeine use: Are they evidenced-based? Semin Fetal Neonatal Med. 2020 Dec;25(6):101177. doi: 10.1016/j.siny.2020.101177. Epub 2020 Nov 4. PMID 33214064
- [Background] Moschino L, Zivanovic S, Hartley C, Trevisanuto D, Baraldi E, Roehr CC. Caffeine in preterm infants: where are we in 2020? ERJ Open Res. 2020 Mar 2;6(1):00330-2019. doi: 10.1183/23120541.00330-2019. eCollection 2020 Jan. PMID 32154294
- [Background] Chen J, Jin L, Chen X. Efficacy and Safety of Different Maintenance Doses of Caffeine Citrate for Treatment of Apnea in Premature Infants: A Systematic Review and Meta-Analysis. Biomed Res Int. 2018 Dec 24;2018:9061234. doi: 10.1155/2018/9061234. eCollection 2018. PMID 30671477
- [Background] Mohammed S, Nour I, Shabaan AE, Shouman B, Abdel-Hady H, Nasef N. High versus low-dose caffeine for apnea of prematurity: a randomized controlled trial. Eur J Pediatr. 2015 Jul;174(7):949-56. doi: 10.1007/s00431-015-2494-8. Epub 2015 Feb 3. PMID 25644724
- [Background] McPherson C, Neil JJ, Tjoeng TH, Pineda R, Inder TE. A pilot randomized trial of high-dose caffeine therapy in preterm infants. Pediatr Res. 2015 Aug;78(2):198-204. doi: 10.1038/pr.2015.72. Epub 2015 Apr 9. PMID 25856169
- [Background] Chavez L, Bancalari E. Caffeine: Some of the Evidence behind Its Use and Abuse in the Preterm Infant. Neonatology. 2022;119(4):428-432. doi: 10.1159/000525267. Epub 2022 Jun 10. PMID 35691280
- [Background] Long JY, Guo HL, He X, Hu YH, Xia Y, Cheng R, Ding XS, Chen F, Xu J. Caffeine for the Pharmacological Treatment of Apnea of Prematurity in the NICU: Dose Selection Conundrum, Therapeutic Drug Monitoring and Genetic Factors. Front Pharmacol. 2021 Jul 26;12:681842. doi: 10.3389/fphar.2021.681842. eCollection 2021. PMID 34381359
- [Derived] Kovacs K, Nagy R, Andreka L, Teutsch B, Szabo M, Varga P, Hegyi P, Harsfalvi P, Acs N, Harmath A, Nador C, Gasparics A. The effect of an additional pre-extubational loading dose of caffeine citrate on mechanically ventilated preterm infants (NEOKOFF trial): Study protocol for a multicenter randomized clinical trial. PLoS One. 2025 Jan 13;20(1):e0315856. doi: 10.1371/journal.pone.0315856. eCollection 2025. PMID 39804861

DOCUMENTS (1):
  • Informed Consent Form (2023-03-14): https://cdn.clinicaltrials.gov/large-docs/83/NCT06401083/ICF_000.pdf